CLINICAL TRIAL: NCT00825630
Title: The Effect of High Dose Citric on PPI (Proton Pump Inhibitors)Induced False Negative H. Pylori UBT Rates
Brief Title: 13-C Urea Breath Test Using BreathID System and PPIs (Proton Pump Inhibitors)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-BID 608
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: HP; UBT; PPI
MeSH Terms: interventions — Lansoprazole; Omeprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lansoprazole (Lanton) (Active Comparator): Patients with H.pylori infection will take one tablet a day of 20 mg Lansoprazole for 14 days orally in the morning
  Interventions: Drug: Lansoprazole (Lanton)
- Omeprazole (Losec) (Active Comparator): Patients with H.pylori infection will take one tablet of 30 mg a day of Omeprazole for 14 days orally in the morning
  Interventions: Drug: Omeprezole (Losec)
- Pantoprazole (Controloc) (Active Comparator): Patients with H.pylori infection will take one tablet a day of 40 mg of Pantoprazole for 14 days orally in the morning
  Interventions: Drug: Pantoprazole(Controloc)
- Esomeprazole(Nexium) (Active Comparator): Patients with H.pylori infection will take one tablet a day of 20 mg Esomeprazole for 14 days orally on the morning
  Interventions: Drug: Esomeprazole (Nexium)

INTERVENTIONS:
Drug: Lansoprazole (Lanton) — Oral administration of Lanzoprazole for 14 days in 25 patients with H.pylori infection
  Other Names: Lanton
  Arms: Lansoprazole (Lanton)
Drug: Omeprezole (Losec) — Oral administration of Omeprazole for 14 days in 25 patients with H.pylori infection
  Other Names: Losec
  Arms: Omeprazole (Losec)
Drug: Pantoprazole(Controloc) — Oral administration of Pantoprazole for 14 days in 25 patients with H.pylori infection
  Other Names: Controloc
  Arms: Pantoprazole (Controloc)
Drug: Esomeprazole (Nexium) — Oral administration of Esomeprazole for 14 days in 25 patients with H.pylori infection
  Other Names: Nexium
  Arms: Esomeprazole(Nexium)

SUMMARY:
Approximately 200 patients with suspected H.pylori will be tested with a 13C-Urea Breath Test (UBT) to ascertain H.pylori positive. 100 H.Pylori positive patients will tested before and after prescribed with one of the four selected Proton Pump Inhibitors (PPIs); 25 patients in each arm. This will provide information on the influence of PPIs on the UBT (Urea Breath Test). The aim of the trial is to observe the effect of different PPIs on the breath test and choose the optimal protocol of when to stop PPI. The hypothesis is that there will be a minimal effect on the UBT while using selected PPIs.

DETAILED DESCRIPTION:
Adult subjects with suspected H pylori infection will be recruited and will undergo a 13C -Urea breath test (including citrica) with the BreathID test device. Those were found positive will undergo selected PPI treatment for 14 days and after 24 or 72 hours from the completion of the two weeks, will undergo a second breath test. Those found to be negative (false negative), will undergo additional breath tests.

* Those subjects that underwent any antibiotic, bismuth or PPI therapy 4 weeks prior to the trial, are to be excluded.
* Furthermore, pregnant or nursing women and subjects with an allergy or sensitivity to one of the tests substrates, will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with H.pylori infection.

Exclusion Criteria:

* Pregnancy,
* Nursing,
* Antibiotic, bismuth or PPI treatment 2 weeks prior to trial,
* Known sensitivity to Urea or citrica.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, MD, Principal Investigator — Sharon Hospital
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Result] Shirin H, Frenkel D, Shevah O, Levine A, Bruck R, Moss SF, Niv Y, Avni Y. Effect of proton pump inhibitors on the continuous real time (13)C-urea breath test. Am J Gastroenterol. 2003 Jan;98(1):46-50. doi: 10.1111/j.1572-0241.2003.07187.x. PMID 12526935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two out-patient clinics in hospitals will enroll subjects
Pre-assignment Details: Size of arms varied due availability of PPI (proton pump inhibitors) and desire to gather more data in most common PPIs.Ethics committees approved additional recruitment.
Groups:
- Lansoprazole (Lanton): Patients with H.pylori infection will take Lanzoprazole orally in the morning (20 mg) for 14 days
- Omeprazole( Losec): Patients with H.pylori infection will take Omeprazole orally in the morning (30mg) for 14 days
- Pantoprazole (Controloc): Patients with H.pylori infection will take Pantoprazole orally in the morning (20mg) for 14 days
- Esomeprazole (Nexium): Patients with H.pylori infection will take Esomeprazole orally in the morning (40mg) for 14 days
Period: Overall Study
Arm/Group | Lansoprazole (Lanton) | Omeprazole( Losec) | Pantoprazole (Controloc) | Esomeprazole (Nexium)
Started | 29 | 62 | 19 | 13
Completed | 29 | 62 | 19 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lansoprazole (Lanton) | Omeprazole( Losec) | Pantoprazole (Controloc) | Esomeprazole (Nexium) | Total
Number analyzed (Participants) | 29 | 62 | 19 | 13 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 55 | 17 | 9 | 107
  >=65 years | 3 | 7 | 2 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.86 (14.67) | 52.48 (13.35) | 51.84 (12.78) | 55.38 (14.84) | 52.46 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 40 | 15 | 7 | 82
  Male | 9 | 22 | 4 | 6 | 41
Region of Enrollment [Number; unit: participants]
  Israel | 29 | 62 | 19 | 13 | 123
H. Pyori Positive [Number; unit: particpants] — Basline particpants include all those with suspected H.pylori infection that are tested with the FDA cleared BreathID 13C urea breath test and are found to be positive, that is DOB (delta over baseline) >=5
  particpants | 29 | 62 | 19 | 13 | 123

OUTCOME MEASURES:

1. Primary Outcome: Urea Breath Test Result (DOB > 5 is Positive)After Different Time Periods From When PPI (Proton Pump Inhibitor) Was Stopped.
Description: Negative value is defined as delta over baseline (DOB) less than 5. The subjects who were positive (DOB>=5) for H.Pylori and after PPI for 10 days repeated a breath with a negative (DOB<5) were considered false negatives. The breath test has been cleared by the FDA in a 510(k) and has > 96% accuracy.
Time Frame: 17 days
Population: Analysis was done on an ITT basis and approximately 25 subjects per group were anticipated in order to obtain a general evaluation of which PPI is will cause the least amount of false negatives.The actual amount of subjects in each group will depend upon the availability of the different PPIs through the course of the study.
Measure: Number; unit: participants
Arm/Group | Lansoprazole (Lanton) | Omeprazole( Losec) | Pantoprazole (Controloc) | Esomeprazole (Nexium)
Number analyzed (Participants) | 29 | 62 | 19 | 13
participants
  False negatives (DOB<5) after 3 days of no PPI | 1 | 3 | 1 | 0
  False negatives (DOB<5) after 1 day of no PPI | 2 | 4 | 2 | 1

ADVERSE EVENTS:
Arm/Group | Lansoprazole (Lanton) | Omeprazole( Losec) | Pantoprazole (Controloc) | Esomeprazole (Nexium)
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/62 | 0/19 | 0/13
Other Adverse Events (participants affected / at risk) | 0/29 | 0/62 | 0/19 | 0/13

LIMITATIONS AND CAVEATS:
It was hard to get people to agree to return for multiple tests within a few days, so the enrollment was difficult

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No